CLINICAL TRIAL: NCT00057057
Title: Randomized Trial of a Telephone Intervention in Heart Failure Patients
Brief Title: Telephone Intervention in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHI 99-074
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure, Congestive; Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Telephone Care

INTERVENTIONS:
Behavioral: Telephone Care

SUMMARY:
In addition to medical treatment for heart failure (HF), a variety of non-pharmacological interventions have been demonstrated to benefit these patients. Some of these include systems for weight monitoring and medication reminders, exercise programs, and individually tailored evaluation and treatment plans with dietitians, social workers, psychologists, and nurse case managers. While many of these approaches have been shown to increase adherence to medication guidelines and result in decreased health care utilization, most rely heavily on a large team of specialized health care providers. It remains unknown whether or not an intervention with a lower intensity of specialized care using sophisticated automated computer tracking and Interactive Voice Response (IVR) techniques can impact the care of HF patients.

DETAILED DESCRIPTION:
Background:

In addition to medical treatment for heart failure (HF), a variety of non-pharmacological interventions have been demonstrated to benefit these patients. Some of these include systems for weight monitoring and medication reminders, exercise programs, and individually tailored evaluation and treatment plans with dietitians, social workers, psychologists, and nurse case managers. While many of these approaches have been shown to increase adherence to medication guidelines and result in decreased health care utilization, most rely heavily on a large team of specialized health care providers. It remains unknown whether or not an intervention with a lower intensity of specialized care using sophisticated automated computer tracking and Interactive Voice Response (IVR) techniques can impact the care of HF patients.

Objectives:

The primary hypothesis of this study is that Heart Failure Telephone Intervention (HearT-I) will decrease hospitalizations and clinic visits in the veteran population with heart failure.

Methods:

The HearT-I intervention consists of three components: 1) computer-initiated medication refill and clinic appointment reminders; 2) IVR access to educational modules; and 3) weekly computer-initiated phone calls with a series of questions regarding weight and symptoms. Four hundred eighty-eight HF patients (NYHA class II-IV) will be randomized to HearT-I intervention vs. usual care. Upon enrollment, all patients will complete questionnaires assessing HF knowledge, behavior, self-efficacy, and perceptions of HF health care, and HF related Quality of Life (Kansas City Cardiomyopathy Questionnaire, KCCQ). Both groups also will receive a digital scale, educational materials, view an educational video about HF and perform a six-minute walk test. We will test the hypothesis that the HearT-I intervention will decrease health care utilization as measured by hospitalizations and unscheduled outpatient visits for HF over one year. Secondary endpoints include KCCQ score, patient satisfaction, adherence to medications, and general knowledge of heart failure and its management.

Status:

Preliminary data analyisis has begun.

ELIGIBILITY:
Inclusion Criteria:

Heart failure NYMA class 2-4, HX of heart failure hospitalization, No COPD, Kansas City Cardiac Questionnaire (Quality of Life)=31-80, 6 minute walk test <450

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Dunlap, MD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States